CLINICAL TRIAL: NCT00467116
Title: A Phase I Study of Erbitux and Gemcitabine With Radiation Therapy for Locally Advanced Pancreas Cancer
Brief Title: PhI Study of Erbitux & Gemcitabine w/Radiation Therapy for Locally Adv. Pancreas Ca
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nipun Merchant, MD, Professor of Surgery and Cancer Biology; Gastrointestinal Surgical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC GI 0466; VU-VICC-GI-0466
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; adenocarcinoma of the pancreas; stage II pancreatic cancer; recurrent pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cetuximab; Gemcitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic Intervention (Experimental)
  Interventions: Biological: cetuximab; Drug: gemcitabine hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Biological: cetuximab — 400mg/m2 initial dose week 1; followed by 250mg/m2/weekly starting week 2 with gemcitabine at fixed dose rate (10 mg/m2/min) + XRT. Cetuximab will start 1 week prior to all other treatment.
  Other Names: Erbitux
Drug: gemcitabine hydrochloride — Dose Level Gemcitabine dose Gemcitabine infusion
  -1 150mg/m2 15 Minutes 0 200mg/m2 20 minutes
  1. 300mg/m2 30 minutes
  2. 400mg/m2 40 minutes
  Other Names: Gemzar
Radiation: radiation therapy — 50.4 Gy, 28 fractions, 5.5 weeks (1.8 Gy/day). A cone down after 45 Gy will be performed to encompass gross disease with a margin of 1-1.5 cm.
  The prescription point will be designated at the intersection of the multiple beams.
  There are no planned interruptions > 3 days.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some find tumor cells and help kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Cetuximab may also stop the growth of tumor cells by blocking blood flow to the tumor. Radiation therapy uses high-energy x-rays to kill tumor cells. Gemcitabine and cetuximab may make tumor cells more sensitive to radiation therapy. Giving gemcitabine together with cetuximab and radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of gemcitabine when given together with cetuximab and radiation therapy in treating patients with locally advanced pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of gemcitabine hydrochloride when administered with cetuximab and radiotherapy in patients with unresectable locally advanced pancreatic or periampullary region cancer.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of gemcitabine hydrochloride.

Patients receive cetuximab IV over 1-2 hours once weekly in weeks 1-7 and gemcitabine hydrochloride IV over 15-40 minutes once weekly in weeks 2-7. Patients also undergo radiotherapy 5 days a week in weeks 2-7. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of gemcitabine hydrochloride until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed for 30 days and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 12-30 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the pancreas (head, body, or tail) or periampullary region, meeting both of the following criteria:

  * Unresectable disease
  * Locally advanced disease
* Measurable or evaluable disease by CT scan or MRI
* No evidence of metastatic disease outside of the planned irradiation field
* ECOG performance status 0-2
* WBC ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8.5 g/dL
* AST and ALT ≤ 5 times upper limit of normal
* Bilirubin ≤ 2.0 mg/dL
* Creatinine ≤ 2.0 mg/dL
* No clinical indication of compromised function of nonirradiated kidney
* No secondary malignancies within the past 5 years except for resected nonmelanoma skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion Criteria:

* No acute hepatitis
* No known HIV infection
* No other active or uncontrolled infection
* No significant history of uncontrolled cardiac disease, including any of the following:

  * Hypertension
  * Unstable angina
  * Myocardial infarction within the past 6 months
  * Congestive heart failure
  * Cardiomyopathy with decreased ejection fraction
* No prior severe infusion reaction to a monoclonal antibody

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to planned field of treatment
* No prior therapy that specifically and directly targets EGFR pathway
* At least 14 days since prior surgery or biopsy
* At least 28 days since prior bypass procedures
* More than 5 years since prior and no other concurrent chemotherapy
* No other concurrent investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2005-10; Primary Completion 2007-08 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Weekly and 4 weeks after last dose of radiation

SECONDARY OUTCOMES:
Dose-limiting toxicity | Weekly and 4 weeks after last dose of radiation
Toxicity | Weekly and 4 weeks after last dose of radiation
Tumor response rate | 4 weeks after last dose of radiation and every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nipun B. Merchant, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States